CLINICAL TRIAL: NCT00005714
Title: Development and Evaluation of Community Asthma Program
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4923; R01HL045293 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2004-08

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To evaluate a community organization approach to promoting asthma management in four neighborhoods in St. Louis with predominantly low income, Black populations.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma prevalence and mortality among Black children exceed levels among whites. Asthma management programs have reduced symptoms, attacks and emergency room usage. However, in 1990 a pattern of underutilization and neglect of care among Black Americans in cases of asthma deaths among Black children indicated the importance of promoting ongoing versus episodic care, reduced exposure to triggers, sensitivity to signs of attacks, attack management, and communication with caregivers, professionals, and teachers. Research in Black communities indicated the importance of informal networks and neighborhood influences, in promoting improved asthma care within low-income Black communities.

The study was part of a demonstration and education initiative "Interventions for Control of Asthma Among Black and Hispanic Children" which was released by the NHLBI in June 1989.

DESIGN NARRATIVE:

Working with an established community agency, Grace Hill Neighborhood Services and its Community Wellness Board, the investigators established Neighborhood Steering Committees to oversee development and implementation of a Neighborhood Asthma Collaboration (NAC) in each neighborhood. The 36-month NAC included (a) promotional campaigns to increase awareness of asthma and its care; (b) Neighborhood Volunteers disseminating leaflets encouraging identification of and continuing care for asthma, and recruiting participants into NAC programs; (c) Neighborhood Volunteers trained as Asthma Advocates to work with asthmatic children and their care-givers to encourage asthma co-management and to conduct management programs in local institutions; (d) an Asthma Management Course offered through community health centers, churches, and other local institutions; and, (e) local school programs including in-service teacher education on asthma management, an asthma program for all students to enhance support for asthmatic children, and school implementation of the Asthma Management Course.

Prior to implementing the NAC, the investigators (a) reviewed, adopted, piloted and revised existing asthma management educational and promotional materials, (b) worked with asthma care providers to gain their involvement in program planning and patient referral to the NAC and (c) adapted procedures from other worksite/community health promotion programs for working with Neighborhood Steering Committees and training Neighborhood Volunteers. General evaluation included (a) surveys of community awareness of and attitudes toward asthma, (b) dissemination and implementation, and (c) pre-post changes in symptoms, attacks, ER visits, and hospitalizations among all child participants in the NAC. These measures as well as kept appointments and serum theophylline levels less than or equal to 5 mg/dl were used in two controlled studies within the NAC to compare (1) children from study neighborhoods with children from socioeconomically comparable neighborhoods, all of whom received care through Children's Hospital of Washington University, and (2) children receiving care through two Centers serving other, socieoeconomically similar neighborhoods.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1990-08; Study Completion 1996-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwin Fisher — Washington University School of Medicine

REFERENCES:
- [Background] Fisher EB Jr, Sussman LK, Arfken C, Harrison D, Munro J, Sykes RK, Sylvia S, Strunk RC. Targeting high risk groups. Neighborhood organization for pediatric asthma management in the Neighborhood Asthma Coalition. Chest. 1994 Oct;106(4 Suppl):248S-259S. doi: 10.1378/chest.106.4_supplement.248s. No abstract available. PMID 7924552
- [Background] Fisher EB Jr, Strunk RC, Sussman LK, Arfken C, Sykes RK, Munro JM, Haywood S, Harrison D, Bascom S. Acceptability and feasibility of a community approach to asthma management: the Neighborhood Asthma Coalition (NAC). J Asthma. 1996;33(6):367-83. doi: 10.3109/02770909609068182. PMID 8968292
- [Background] Munro JF, Haire-Joshu D, Fisher EB, Wedner HJ. Articulation of asthma and its care among low-income emergency care recipients. J Asthma. 1996;33(5):313-25. doi: 10.3109/02770909609055372. PMID 8827938